CLINICAL TRIAL: NCT00332319
Title: See Detailed Description
Brief Title: Effects Of GW679769 On Bladder Nerve Function And Symptoms Of Overactive Bladder In Spinal Cord Injury Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NKB104846
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2011-03

CONDITIONS: Incontinence, Urinary and Urinary Bladder, Overactive; Overactive Bladder
Keywords: spinal cord injury; urgency; Overactive bladder; neurogenic; neurometry; frequency; urge incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Spinal Cord Injuries; Urinary Incontinence, Urge | interventions — casopitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW679769

SUMMARY:
This is a two-part study in which Part A will assess the effects of GW679769 after 1 dose on the function of the nerves that supply the bladder. The technique for measuring the nerves function is called Neurometry. Part B will assess the effect of repeat doses of GW679769 on the bladder nerve function. Part B will also assess the effects of the drug on overactive bladder symptoms using a three-day patient diary.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study to evaluate the effects of GW679769 on Current Perception Threshold (CPT) following a single 150 mg dose (Part A) and to evaluate the effect of CPT and symptoms of overactive bladder following 28 days of repeat dosing with 120 mg GW679769 administered once daily (Part B) in patients with neurogenic bladder due to incomplete spinal cord injury

ELIGIBILITY:
Inclusion criteria:

* Spinal cord injury patients with overactive bladder symptoms including urge incontinence, urgency, frequency and night-time urination but without bladder related pain.
* The injury must be above S1-3

Exclusion criteria:

* Spinal cord injury suffered within 6 months.
* History of interstitial cystitis, radiation cystitis, pelvic irradiation, or myocardial infarction with 1 year prior to screening.
* Pregnant or nursing females.
* Patients who have had hypersensitivity to lidocaine.
* Patients who are taking oral corticosteroids.
* Patients with active peptic ulcer disease (PUD) and/or history of PUD of an unknown etiology.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Change in bladder nerve activity assessed by neurometry before and after a single dose of GW679769 and placebo (part A) and after 28 days of drug or placebo treatment (part B).

SECONDARY OUTCOMES:
Improvement of OAB symptoms (incontinence, frequency of urination, reduction in urgency, decrease in night-time urination episodes).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania